CLINICAL TRIAL: NCT02926742
Title: Submassive Pulmonary Embolism Experience With EKOS
Acronym: SPEEK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Krishna Mannava, MD, FACS, RPVI (Other)
Collaborators: EKOS Corporation (Industry)
Responsible Party: Sponsor-Investigator, Krishna Mannava, MD, FACS, RPVI, Krishna Mannava, MD, FACS, RPVI, Fairfield Medical Center
Organization: Fairfield Medical Center (Other)
Other Study IDs: FMCspeekEKOSstudy
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Thrombolytic Therapy; Thrombolysis; Mechanical Thrombolysis; Pulmonary Embolism
Keywords: Thrombolysis; Ultrasound Thrombolysis; Pulmonary Embolism; Saddle PE; Submassive PE; Massive PE; Bilateral PE
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: EkoSonic Endovascular System — Ultrasound catheter-directed thrombolysis.

SUMMARY:
This single site study evaluates the efficacy of ultrasound accelerated thrombolysis using EKOS Endovascular Device with a standard infusion of thrombolytics for treatment of PE

DETAILED DESCRIPTION:
Previous clinical trials examining thrombolytics used to treat Acute Submassive PE, many times will use fixed dose and duration. Little research has been conducted on the physiologic implication of resolution of symptoms. It seems reasonable, that symptomatic relief results from some degree of hemodynamic normalization. This study will seek to examine the extent to which the hemodynamic impairment is normalized from a thrombolytic treatment protocol with an endpoint of therapy determined as resolution of presenting symptoms. Treatment plans will utilize the MBS (Modified Borg Scale) score to help evaluate and measure outcome-based care, quantifying shortness of breath.

ELIGIBILITY:
Inclusion Criteria:

1. Acute symptomatic PE confirmed by CT, with filling defect in at least one main or segmental pulmonary artery.
2. RV dysfunction as evidenced by RV/LV ratio > 0.9 on echo
3. Ability to give informed consent or Legally Authorized Representative (LAR) is able to give consent
4. PE symptom duration < 21 days
5. Age >18 years
6. And, a MBS baseline measurement above 3 plus at least one of the following: O2 sat < 90% RA, or inability to maintain a HR <100, or inability to maintain a Systolic Bp > 100. Whichever measurement is chosen for inclusion criteria in addition to the MBS will also be used in determination of therapeutic endpoint (i.e. O2 Sat., HR<100 or BP >100)..

Exclusion Criteria:

1. Stroke or transient ischemic attack (TIA), head trauma, or other active intracranial or intraspinal disease within one year
2. Recent (within one month) or active bleeding from a major organ
3. Hemoglobin (Hgb) < 8.0
4. Platelets < 60 thousand/µL
5. Major surgery within seven days
6. Clinician deems high-risk for catastrophic bleeding
7. History of heparin-induced thrombocytopenia (HIT)
8. Pregnancy
9. Catheter-based pharmacomechanical treatment for pulmonary embolism within 3 days of study enrollment
10. Systolic blood pressure less than 80 mm Hg despite vasopressor or inotropic support
11. Cardiac arrest (including pulseless electrical activity and asystole) requiring active cardiopulmonary resuscitation (CPR)
12. Evidence of irreversible neurological compromise
13. Life expectancy < 30 days
14. Use of thrombolytics or glycoprotein IIb/IIIa antagonists within 3 days prior to inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital setting. Volunteers meeting the inclusion/ exclusion criteria who are patients of Fairfield Medical Center located in Lancaster, Oho
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Reduction of RV dysfunction | 48 hours post catheter removal
  Reduction of RV dysfunction as evidenced by a reduction in RVSP and or a reduction in RV/LV ratio measured by echo at baseline and again at 48 ±6 hours post EKOS catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Lisa K Stevens, MSN, Study Director — Fairfield Medical Center; Krishna Mannava, MD, Principal Investigator — Fairfield Medical Center
Locations (1):
- Fairfield Medical Center, Lancaster, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified individual study participant data will be made available 6 months after study completion. This data to include all primary and secondary outcome measures.